CLINICAL TRIAL: NCT04171297
Title: Ultrasound Evaluation of the Pelvis Using the International Deep Endometriosis Analysis (IDEA) Terminology in Women with Suspected Endometriosis Scheduled for Laparoscopic Surgery - IDEA 1 Study
Brief Title: Ultrasound Evaluation of the Pelvis in Women with Suspected Endometriosis Scheduled for Laparoscopic Surgery
Acronym: IDEA1
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University of Sydney (Other); University of Cagliari (Other)
Responsible Party: Sponsor
Other Study IDs: S63056
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Gynecologic Disease; Endometriosis; Endometriosis, Rectum; Endometriosis of Colon; Endometriosis of Vagina; Endometriosis Rectovaginal Septum; Endometriosis of Bladder; Surgery
MeSH Terms: conditions — Genital Diseases, Female; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Ultrasound evaluation of DE — To evaluate diagnostic accuracy of ultrasound for the presence of deep endometriosis.

SUMMARY:
An international multicenter observation study to evaluate the diagnostic accuracy and predictive value of ultrasound using the IDEA terminology in the detection of deep endometriosis in women scheduled for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for radical laparoscopic endometriosis surgery

Exclusion Criteria:

* <18 years
* >45 years
* (suspected) Pelvic malignancy for example gynecological, intestinal or urological malignancy
* Premenarche
* Menopause
* Pregnancy
* Patients refusal for radical surgery (for example refusal for bowel resection/temporary stoma)
* Surgery performed more than 1 year after ultrasound scan
* Patients refusal to participate to the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with suspected endometriosis scheduled for laparoscopic surgery.
Sampling Method: Probability Sample
Enrollment: 1866 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Presence of deep endometriosis | 1 year
  The primary objective is to assess the diagnostic value of the ultrasound features in the diagnosis of deep endometriosis. The endpoints are the univariable diagnostic accuracies of ultrasound features (defined by the IDEA consensus statement) for the presence of deep endometriosis at any location: anterior compartment (i.e. bladder and its specific location) or posterior compartment (i.e. rectovaginal septum, uterosacral ligaments, torus uterinus, vaginal fornix and bowel involvement). All recruited patients are included in this analysis. The reference standard for this objective is whether there is deep endometriosis (at any location) or not (binary outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Timmerman, MD, PhD, Principal Investigator — UZ Leuven
Locations (3):
- Sydney Medical School Nepean, Sydney, Australia
- UZLeuven, Leuven, Belgium
- University of Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No